CLINICAL TRIAL: NCT06651515
Title: A Phase 1/2 Adaptive Dose Study to Evaluate the Safety and Efficacy of SR-02 Pancreatic Endocrine Cell Clusters Implanted in the Omentum of Adults With Type 1 Diabetes
Brief Title: A Study of the Safety and Efficacy of Pancreatic Endocrine Cell Clusters Implanted Into the Omentum of Type 1 Diabetes Patients With Severe Hypoglycemia
Acronym: SUGR
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study is being withdrawn for business reasons
Sponsor: Seraxis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR-02-201
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus Type 1
Keywords: severe hypoglycemia; diabetes mellitus; endocrine system diseases; glucose metabolism disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SR-02 Allogeneic pancreatic endocrine cell clusters (Experimental)
  Interventions: Biological: Allogeneic Pancreatic Endocrine Cell Clusters

INTERVENTIONS:
Biological: Allogeneic Pancreatic Endocrine Cell Clusters — Allogeneic Pancreatic Endocrine Cell Clusters

SUMMARY:
This study will evaluate the safety, efficacy and durability of SR-02 administered to the omentum of patients of Type 1 diabetes with severe recurrent hypoglycemia. The study will also help establish the optimal treatment dose. Although this study is open to patients with all HLA or blood types, immunosuppression to prevent rejection will be required in this first in human study.

ELIGIBILITY:
Key Inclusion Criteria

* Adult 18 to 65 years with a clinical history of T1D
* Diagnosis of T1D at <40 years of age
* insulin dependence for ≥5 years at pre-screening
* Recurrent severe hypoglycemia
* Willingness to use continuous glucose monitoring

Key Exclusion Criteria

* Use of anti-diabetic agent other than insulin(s) or insulin analog(s) within 3 months of Screening
* Weight loss medication(s) within 3 months of Screening

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety and tolerability based on the percentage and relatedness of all treatment emergent adverse events and serious adverse events (TEAEs and SAEs) | day 35 through day 365
The effect on endogenous insulin secretion as assessed by 90-minute MMTT-stimulated C-peptide >0.5 ng/ml (>0.17 nmol/L) | 90 day intervals through day 365

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No